CLINICAL TRIAL: NCT00756639
Title: Prophylactic Cranial Irradiation (PCI) for Patients With Small Cell Carcinoma of the Urothelium
Brief Title: Prophylactic Cranial Irradiation (PCI) for Small Cell Carcinoma of the Urothelium
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0933; NCI-2012-01675 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-09-18; First posted 2008-09-22 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Bladder Cancer
Keywords: small cell carcinoma of the bladder; urothelial carcinoma; genitourinary bladder; urothelium; bladder; bladder cancer; prophylactic cranial irradiation; PCI; brain metastasis; genitourinary; radiation; TCC; adenocarcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell; Brain Neoplasms; Adenocarcinoma | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- Radiation (Experimental): Prophylactic cranial irradiation (PCI) treatments to be started within 4 months after the end of chemotherapy or surgery to a total dose of 30 Gy, given at 2 Gy per fraction, 5 days per week for 3 weeks. On the first day of each week of therapy, a brain X-ray will done to see if the radiation is being given to the best area.
  Interventions: Radiation: Prophylactic Cranial Irradiation (PCI); Other: Brain X-ray

INTERVENTIONS:
Radiation: Prophylactic Cranial Irradiation (PCI) — Prophylactic cranial irradiation (PCI) treatments to be started within 4 months after the end of chemotherapy or surgery to a total dose of 30 Gy, given at 2 Gy per fraction, 5 days per week for 3 weeks.
  Other Names: Whole Brain Radiation; Prophylactic cranial irradiation; PCI
Other: Brain X-ray — On the first day of each week of therapy, a brain X-ray will done to see if the radiation is being given to the best area.
  Other Names: X-ray

SUMMARY:
The goal of this clinical research study is to learn if whole brain radiation can lower the chances of developing brain tumors in patients with small cell carcinoma of the urinary tract, including the bladder. The safety of whole brain radiation will also be studied.

DETAILED DESCRIPTION:
Pregnancy Test:

Women who are able to have children must have a negative urine pregnancy test to be eligible for this study.

MRI/CT Scans:

Within six (6) weeks before having whole brain radiation, you will have a magnetic resonance imaging (MRI) or a computed tomography (CT) scan of your brain to check if brain tumors have developed.

Simulation Visit:

Before the radiation therapy begins, you will have a "simulation visit" to plan for the radiation therapy. During this session, you will be fitted to a plastic mask to hold your head still during radiation. The mask is made of a material called "thermoplastic" that becomes soft when it is placed in warm water. While this plastic is soft, it will be pulled over your face to make a mold. When the plastic cools down, it will harden again and the mask will be completed. After the mask is made, a CT scan of your head will be done for treatment planning.

Radiation Therapy:

You will begin radiation within 1 week after the simulation visit. You will have radiation visits Monday through Friday for 3 weeks (15 total therapy visits). Each therapy session will last about 15 minutes. It will take the study staff about 10 minutes to position you on the table and put the mask on. The radiation will be given over 2-3 minutes.

On the first day of each week of therapy, you will have a brain X-ray to see if the radiation is being given to the best area.

Follow-Up:

After the radiation therapy, you will have an MRI or a CT scan of the brain every 6 months for 1 year and then every year for 5 years to check the status of the disease. More frequent scans will be performed if your doctor thinks they are needed. You will also complete a written mental status exam with your doctor every 3-6 months for 2 years and then every year for 5 years. The exam will have a series of tests to check your memory and ability to follow instructions. The test will take about 15 minutes to complete.

Length of Study:

You may remain on study for as long as you are benefitting. You will be taken off study if your disease gets worse or if intolerable side effects occur.

This is an investigational study. The use of radiation to check for brain tumors before they have formed is investigational.

Up to 30 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven small cell carcinoma of the bladder, or elsewhere along the urothelium, which is locally advanced or metastatic (i.e. > or = cT3b, > or = pT3b, N+, or M+) at the time of presentation or cystectomy who have been treated with chemotherapy.
2. Patients must have had a response to chemotherapy, which the investigator feels is likely to resulting systemic control of the cancer. In most instances, this would reflect a major response (i.e. > or = 90% reduction of tumor), though a lower percentage may be acceptable if the investigator feels the residual reflects another component, such as transitional cell carcinoma (TCC). Dr Arlene Siefker-Radtke will serve as the final arbiter when questions regarding response arise.
3. Since small cell tumors of the bladder are often associated with other variant histology including TCC and adenocarcinoma, the presence of variant histology will be allowed.
4. Patients must be > or = 18 years of age.
5. Patients may be on other trials (either here at M.D. Anderson Cancer Center or at an outside institution) as long as the other eligibility criteria are met.
6. Patients must not have any evidence of progressive disease at the time of study entry.
7. Patients must have an MRI or CT of the head showing no CNS metastases within 6 weeks of study entry.
8. Patients must have adequate physiologic reserves as evidenced by: a) Zubrod Performance Status (PS) of < or = 2; b) Adequate bone marrow reserves as evidenced by ANC > 1000, and platelet count > 75,000. Supranormal values judged to be of benign or inconsequential etiology will be acceptable.
9. Patients must be enrolled within 6 months of completing chemotherapy or after surgery of the primary site. Any acute/subacute > or = grade 3 toxicities from the chemotherapy must be resolved to < or = grade 2 at the time of study entry. It is suggested that patients undergo prophylactic cranial irradiation as a soon as they have recovered from chemotherapy or surgery, at a minimum of 2 weeks, and up to 6 months following chemotherapy or surgery.

Exclusion Criteria:

1. Patients with CNS metastasis at presentation will not be eligible.
2. History of TIA or stroke within 6 months of study entry.
3. Prior cranial irradiation.
4. Pregnant women will not be eligible; women of childbearing potential must have a negative pregnancy test before starting therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-07-21 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Brain Metastasis Free Survival | At 1 Year
  Primary outcome for this trial is the rate of development of brain metastasis by 12 months following start of treatment. A "success" defined as a patient not developing brain metastasis by 12 months following start of treatment. After radiation therapy, participant has an MRI or a CT scan of the brain every 6 months for 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Seungtaek Choi, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org